CLINICAL TRIAL: NCT02094456
Title: Prophylactic Elective Clipping of Colonic Diverticula in Patients Who Have Had Sustained Lower Gastrointestinal Haemorrhage
Brief Title: Prophylactic Elective Clipping of Colonic Diverticula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14/LO/0032
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2016-04

CONDITIONS: Diverticular Disease
Keywords: diverticular disease; diverticular bleeding; endoscopic clipping; endoscopy; lower gastrointestinal bleeding
MeSH Terms: conditions — Diverticular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoscopic clipping of diverticula (Experimental): Endoscopic clipping of diverticula Follow-up colonoscopy
  Interventions: Procedure: Endoscopic clipping of diverticula; Procedure: Follow-up colonoscopy

INTERVENTIONS:
Procedure: Endoscopic clipping of diverticula — Colonoscopy with identification of each individual colonic diverticula and endoscopic clipping.
Procedure: Follow-up colonoscopy — Patients will undergo a repeat colonoscopy 6 months after endoscopic clipping procedure.

SUMMARY:
Diverticular bleeding is the most common cause of acute lower gastrointestinal bleeding (LGIB) in Western populations. Although self-limited in 85% of cases, some patients may require hospitalization with blood transfusion and emergent intervention, with significant associated morbidity and mortality. Up to 25% of patients with an initial bleeding episode will have subsequent episodes.

Diverticula form at weak points along the colon wall, where the vasa recta enter the circular muscle layer of the colon. Diverticular bleeding is attributed to thinning of the blood vessels as they cross over the dome of a diverticulum. Endoscopic clipping of actively bleeding colonic diverticula has been recognized as a safe and effective treatment for acute LGIB since the mid1990s. Patients selected would have had previous colonoscopy to exclude other causes of bleeding (e.g. angiodysplasia, colorectal cancer).

The investigators propose prophylactic elective endoscopic diverticular clipping in patients who have had at least 1 episode of acute LGIB requiring hospitalization. This would involve applying endoscopic clips to the base of every diverticula in a patient's colon, such that any bleeding source would effectively be excluded. The investigators would later reevaluate patients for colonoscopic appearance of diverticula to assess their diverticular disease.

The investigators hypothesize that patients undergoing endoscopic diverticular clipping will not have repeat episodes of bleeding.

DETAILED DESCRIPTION:
1.0 BACKGROUND AND HYPOTHESES

The investigators aim to prophylactically clip all colonic diverticula in patients who have experienced at least 1 episode of diverticular bleeding requiring hospitalization, but without definitive procedure (i.e., total colectomy or localization with embolization or clipping). The investigators' objective is to prevent future episodes of colonic bleeding from the diverticula, so as to avoid morbidity and possible mortality.

The investigators hypothesize that those patients undergoing secondary prophylaxis through diverticular clipping will experience no further episodes of diverticular bleeding.

2.0 OBJECTIVES AND PURPOSE

Diverticular bleeding is the most common cause of acute lower gastrointestinal bleeding (LGIB) in Western populations. Although self-limited in 85% of cases, some patients may require hospitalization with blood transfusion and emergent intervention, with significant associated morbidity and mortality. Up to 25% of patients with an initial bleeding episode will have subsequent episodes.

Diverticula form at weak points along the colon wall, where the vasa recta enter the circular muscle layer of the colon. Diverticular bleeding is attributed to thinning of the blood vessels as they cross over the dome of a diverticulum. Endoscopic clipping of actively bleeding colonic diverticula has been recognized as a safe and effective treatment for acute LGIB since the mid-1990s. Patients selected would have had previous colonoscopy to exclude other causes of bleeding (e.g. angiodysplasia, colorectal cancer).

The investigators propose prophylactic elective endoscopic diverticular clipping in patients who have had at least 1 episode of acute LGIB requiring hospitalization. This would involve applying endoscopic clips to the base of every diverticula in a patient's colon, such that any bleeding source would effectively be excluded. The investigators would later re-evaluate patients for colonoscopic appearance of diverticula, as there is some suggestion that diverticula may resolve after such management.

3.0 STUDY DESIGN

The investigators propose a prospective feasibility study of outpatients who have previously been hospitalized with at least one episode of diverticular bleeding. Diverticular disease will have been confirmed by previous colonoscopy to assess the extent of diverticular disease. Consecutive patients at follow-up outpatient appointments will be approached with a Patient Information Sheet. On follow-up appointment they will be recruited and enrolled for endoscopic clipping of colonic diverticula.

The procedure itself will be similar to a screening colonoscopy. As outpatients, patients will take bowel preparation. Colonoscopy will occur with sedation only, including fentanyl and midazolam per protocol. Individual colonic diverticula will be clipped to exclude the bleeding source.

Twenty-four (24) patients will be enrolled for diverticular clipping. These patients will be followed prospectively for 2 years for repeat bleeding episodes. Follow-up will consist of telephone calls every 6 months by the study team. In addition, patients will be scheduled for repeat colonoscopy to assess their diverticular disease 6 months after clipping of colonic diverticula.

4.0 SELECTION AND WITHDRAWAL OF SUBJECTS Currently, patients admitted with complications of diverticular disease are seen in Diverticular Disease clinic for follow-up. Consecutive patients will be selected from this patient population.

Patients may withdrawal from the study at any time, including during the colonoscopy with clipping of diverticula.

5.0 DATA COLLECTION AND MONITORING

Data collection will take place on a specially created case report form (See case report form version 1.2). Case report forms will be stored in a locked office in the Department of Colorectal Surgery accessible only to the study team. Data will be entered into an excel spreadsheet. The spreadsheet will be kept on a password protected NHS desktop in a locked office in the Department of Colorectal Surgery.

6.0 STATISTICAL CONSIDERATIONS

As this is a feasibility study, recruited patients will be study prospectively. Any analysis will include all patients enrolled. There will be no control group or randomization at this time.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they have been hospitalized at least once with diverticular bleeding.

Exclusion Criteria:

* Patients who had a definitive procedure to stop diverticular bleeding, including colectomy or angiography with embolization.
* Patients who are considered too high risk for colonoscopy or bowel preparation. There will be no exclusion criteria based on age. Rather, patients will be individually evaluated and judged for frailty.
* Patients on anticoagulant agents that may not be stopped for colonoscopy.
* Patients without colonic diverticula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be episodes of recurrent bleeding requiring hospitalization. | 12 months
  Postprocedure, patients will follow-up every 6 months either in Diverticular Disease clinic or via telephone checkup. These visits will ascertain whether patients have had recurrent bleeding episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Amyn Haji, MSc MD FRCS, Principal Investigator — King's College Hospital NHS Trust; Charlotte Kvasnovsky, MD MPH, Study Director — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, United Kingdom